CLINICAL TRIAL: NCT06858839
Title: A Phase 3 Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy, Safety, and Tolerability of Maridebart Cafraglutide in Adult Participants Without Type 2 Diabetes Mellitus Who Have Obesity or Are Overweight
Brief Title: Evaluation of Maridebart Cafraglutide in Adult Participants Without Type 2 Diabetes Mellitus Who Have Obesity or Are Overweight
Acronym: MARITIME-1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20210181; 2024-515524-36 (EudraCT Number)
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Obesity
Keywords: Overweight; BMI; Body weight; Maridebart cafraglutide; Chronic weight management; MariTide
MeSH Terms: conditions — Obesity; Overweight; Body Weight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Maridebart Cafraglutide High Dose (Experimental): Participants will receive maridebart cafraglutide high dose subcutaneously (SC) for 72 weeks.
  Interventions: Drug: Maridebart Cafraglutide
- Maridebart Cafraglutide Medium Dose (Experimental): Participants will receive maridebart cafraglutide medium dose SC for 72 weeks.
  Interventions: Drug: Maridebart Cafraglutide
- Maridebart Cafraglutide Low Dose (Experimental): Participants will receive maridebart cafraglutide low dose SC for 72 weeks.
  Interventions: Drug: Maridebart Cafraglutide
- Placebo (Placebo Comparator): Participants will receive placebo SC for 72 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Maridebart Cafraglutide — Maridebart cafraglutide will be administered SC.
  Other Names: AMG 133; MariTide
  Arms: Maridebart Cafraglutide High Dose; Maridebart Cafraglutide Low Dose; Maridebart Cafraglutide Medium Dose
Drug: Placebo — Placebo will be administered SC.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to demonstrate that maridebart cafraglutide is superior to placebo for percent change in body weight.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Body mass index ≥ 30 kg/m2 or ≥27 kg/m² to < 30 kg/m2 with at least 1 of the following weight-related comorbidities: hypertension, dyslipidemia, history of obstructive sleep apnea, history of cardiovascular disease, history of metabolic dysfunction-associated steatotic liver disease (MASLD) or Metabolic Dysfunction-Associated Steatohepatitis (MASH).
* History of at least 1 self-reported unsuccessful attempt at weight loss by diet and exercise.

Exclusion Criteria:

* Type 1 or Typ2 diabetes mellitus.
* Obesity induced by other endocrinologic disorders.
* Self-reported change in body weight > 5 kg within 90 days before screening.
* Family (first-degree relative[s]) or personal history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2.
* History of chronic pancreatitis or history of acute pancreatitis within 180 days before screening.
* History of unstable major depressive disorder (MDD) or other severe psychiatric disorder within 2 years before screening.
* Lifetime history of suicide attempt.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3853 (Actual)
Dates: Start 2025-03-12 (Actual); Primary Completion 2027-01-21 (Estimated); Study Completion 2027-04-16 (Estimated)

PRIMARY OUTCOMES:
Percent Change From Baseline in Body Weight at Week 72 | Baseline and Week 72

SECONDARY OUTCOMES:
Change From Baseline in Waist Circumference at Week 72 | Baseline and Week 72
Participant achieving ≥ 5% reduction in body weight from baseline at week 72 | Week 72
Participant achieving ≥ 10% reduction in body weight from baseline at week 72 | Week 72
Participant achieving ≥ 15% reduction in body weight from baseline at week 72 | Week 72
Participant achieving ≥ 20% reduction in body weight from baseline at week 72 | Week 72
Change From Baseline in Systolic Blood Pressure (SBP) at Week 72 | Baseline and Week 72
Percent Change From Baseline in Fasting Triglycerides at Week 72 | Baseline and Week 72
Change From Baseline in Fasting Glucose at Week 72 | Baseline and Week 72
Change From Baseline in the Impact of Weight on Quality of Life-Lite Clinical Trials Version (IWQOL-Lite-CT) Physical Function Composite Score at Week 72 | Baseline and Week 72
  The IWQOL-Lite-CT is a 20-item questionnaire designed to assess the impact of weight on quality of life in clinical trials. Items are scored on a 5-point Likert scale, with raw scores transformed to a 0-100 scale, where higher scores indicate better quality of life and less weight-related impact.
Change From Baseline in Body Weight at Week 72 | Baseline and Week 72
Change From Baseline in Body Mass Index (BMI) at Week 72 | Baseline and Week 72
Change From Baseline in Hemoglobin A1c at Week 72 | Baseline and Week 72
Percent Change From Baseline in Fasting Insulin at Week 72 | Baseline and Week 72
Change From Baseline in Glycemic Status at Week 72 | Baseline and Week 72
Percent Change From Baseline in Fasting Lipid Parameters at Week 72 | Baseline and Week 72
  Lipid parameters include: total cholesterol, non-high-density lipoprotein cholesterol (non-HDL-C), low-density lipoprotein cholesterol (LDL-C), very-low-density lipoprotein cholesterol (VLDL-C), and high-density lipoprotein cholesterol (HDL-C).
Change From Baseline in Diastolic Blood Pressure (DBP) at Week 72 | Baseline and Week 72
Percent Change From Baseline in High-sensitivity C-reactive Protein (hs-CRP) at Week 72 | Baseline and Week 72
Change From Baseline in Short Form 36 Health Survey Version 2 (SF-36v2) Acute Physical Function Domain Score at Week 72 | Baseline and Week 72
  The SF-36v2 Acute Physical Function domain score measures an individual's ability to perform daily physical activities, such as walking and climbing stairs, over the past week. It includes 10 items scored on a 3-point Likert scale, with raw scores transformed to a 0-100 scale. Higher scores indicate better physical functioning and fewer limitations due to physical health.
Number of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | Up to approximately 88 weeks
Plasma Concentration of Maridebart Cafraglutide at Week 72 | Week 72

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (242):
- United States (73):
  - Pinnacle Research Group LLC, Anniston, Alabama
  - Alliance For Multispecialty Research - Daphne, Daphne, Alabama
  - Alliance for Multispecialty Research Mobile, Mobile, Alabama
  - Avacare Foothills Research Center, Phoenix, Arizona
  - Ark Clinical Research- Tustin, Fountain Valley, California
  - Long Beach Clinical Trials Services Inc, Long Beach, California
  - Ark Clinical Research- Long Beach, Long Beach, California
  - Catalina Research Institute, Montclair, California
  - Artemis Institute for Clinical Research, Riverside, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Apex Clinical Research, San Diego, California
  - Southern California Clinical Research, Santa Ana, California
  - Diablo Clinical Research, Walnut Creek, California
  - Yale School of Medicine, New Haven, Connecticut
  - Chase Medical Research LLC, Waterbury, Connecticut
  - Indago Research and Health Center, Hialeah, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Clinical Neuroscience Solutions - Jacksonville, Jacksonville, Florida
  - South Florida Wellness and Clinical Research Institute, Margate, Florida
  - Optimus U Corporation, Miami, Florida
  - Research Institute of South Florida, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Clinical Neuroscience Solutions - Orlando, Orlando, Florida
  - Combined Research Orlando Phase I IV, Orlando, Florida
  - Florida Institute for Clinical Research, Orlando, Florida
  - Encore Medical Research of Weston LLC, Weston, Florida
  - Center for Advanced Research and Education, Gainesville, Georgia
  - Rophe Adult and Pediatric Medicine/Sky Clinical Research Network Group, Union City, Georgia
  - East-West Medical Research, Honolulu, Hawaii
  - Solaris Clinical Research, Meridian, Idaho
  - Flourish Research - Great Lakes Clinical Trials, Chicago, Illinois
  - Endeavor Health Medical Group - Endocrinology and Diabetes- Skokie, Skokie, Illinois
  - Evanston Premier Healthcare Research LLC, Skokie, Illinois
  - Alliance for Multispecialty Research Newton, Newton, Kansas
  - Louisville Metabolic and Atherosclerosis Research Center, Louisville, Kentucky
  - Velocity Clinical Research - Baton Rouge, Baton Rouge, Louisiana
  - Tandem Clinical Research - Marrero, Marrero, Louisiana
  - Headlands Research - Detroit, Southfield, Michigan
  - Prime Health and Wellness Sky Clinical Research Network Group, Fayette, Mississippi
  - Alliance for Multispecialty Research - Kansas City, Kansas City, Missouri
  - Palm Research Center Inc, Las Vegas, Nevada
  - Vector Clinical Trials, Las Vegas, Nevada
  - Rochester Clinical Research, Rochester, New York
  - Velocity Clinical Research- Binghamton, Vestal, New York
  - Accellacare of Hickory, Hickory, North Carolina
  - Carolina Research Center Inc, Shelby, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Clinical Trial Investigator Clinical Research Center, Cincinnati, Ohio
  - Velocity Clinical Research - Cincinnati, Cincinnati, Ohio
  - Alliance for Multispecialty Research - Norman, Norman, Oklahoma
  - Capital Area Research LLC, Newport, Pennsylvania
  - Velocity Clinical Research - Providence, East Greenwich, Rhode Island
  - Tribe Clinical Research LLC Dba Mountain View Clinical Research, Greenville, South Carolina
  - New Phase Research and Development, Knoxville, Tennessee
  - Accellacare US Inc., d/b/a Accellacare of Knoxville, Knoxville, Tennessee
  - Elligo Clinical Research Center, Austin, Texas
  - Cedar Health Research, LLC, Dallas, Texas
  - Epic Medical Research - Texas, DeSoto, Texas
  - Great Lakes Research Institute El Paso Research, El Paso, Texas
  - Cedar Health Research, LLC, Euless, Texas
  - Juno Research LLC, Houston, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Southern Endocrinology Associates PA, Mesquite, Texas
  - Great Lakes Research Institute - McAllen Research, Pharr, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - Sugar Lakes Family Practice, Sugar Land, Texas
  - Pantheon Clinical Research, Bountiful, Utah
  - Alliance for Multispecialty Research Layton Research Center, Layton, Utah
  - Chrysalis Clinical Research, LLC, St. George, Utah
  - Washington Center for Weight Management and Research, Inc, Arlington, Virginia
  - Health Research of Hampton Roads, Newport News, Virginia
  - Selma Medical Associates, Winchester, Virginia
  - Allegiance Research Specialists, Milwaukee, Wisconsin
- Argentina (8):
  - Cedic - Centro de Investigacion Clinica, CABA, Buenos Aires
  - Centro Medico Viamonte, CABA, Buenos Aires
  - Cemedic Centro de Especialidades Medicas, CABA, Buenos Aires
  - Centro Medico Dra Laura Maffei Investigacion Clinica Aplicada, CABA, Buenos Aires
  - Consultorios Medicos Dr Besada, CABA, Buenos Aires
  - Fundacion Respirar, CABA, Buenos Aires
  - Cinme - Centro de Investigaciones Metabolicas, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Ciprec - Centro de Investigacion y Prevencion Cardiovascular, Ciudad Autonoma de Buenos Aires, Buenos Aires
- Australia (11):
  - Emeritus Research Sydney, Botany, New South Wales
  - Novatrials, Charlestown, New South Wales
  - Canopy Clinical Sutherland, Miranda, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Canopy Clinical Wollongong, Wollongong, New South Wales
  - Logan Hospital, Meadowbrook, Queensland
  - Fusion Clinical Research, Norwood, South Australia
  - Southern Adelaide Diabetes and Endocrine Services, Oaklands Park, South Australia
  - Emeritus Research Camberwell, Camberwell, Victoria
  - Austin Health, Heidelberg Repatriation Hospital, Heidelberg West, Victoria
  - Canopy Clinical Altona North, North Altona, Victoria
- Belgium (7):
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - Algemeen Ziekenhuis Groeninge - Campus Kennedylaan, Kortrijk
  - Universitair Ziekenhuis Leuven - Campus Gasthuisberg, Leuven
  - Centre Hospitalier Universitaire de Liege - Sart Tilman, Liège
  - Algemeen Ziekenhuis Sint-Maarten, Mechelen
  - Centres Hospitaliers Universitaires HELORA - Hôpital de Mons - Site Constantinople, Mons
- Canada (12):
  - tlc Diabetes and Endocrinology, Surrey, British Columbia
  - Wharton Medical Clinic, Hamilton, Ontario
  - North York Diagnostic and Cardiac Centre, North York, Ontario
  - Centricity Research Oshawa Multispecialty, Oshawa, Ontario
  - Heart Health Institute Research Incorporated, Scarborough Village, Ontario
  - Curans Heart Center, Thunder Bay, Ontario
  - Centricity Research Toronto, Toronto, Ontario
  - Diabetes Heart Research Centre, Toronto, Ontario
  - Ecogene-21, Chicoutimi, Quebec
  - Institut Universitaire de cardiologie et de pneumologie de Quebec, Québec, Quebec
  - CardioVasc HR Incorporated, Saint-Jean-sur-Richelieu, Quebec
  - Centre de Medecine Metabolique de Lanaudiere, Terrebonne, Quebec
- Czechia (11):
  - Medicus Services sro, Brandýs nad Labem
  - Fakultni nemocnice Brno, Brno
  - Endohope Havirov sro, Havířov
  - PreventaMed sro, Olomouc
  - CCR Ostrava sro, Ostrava
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Ob klinika as, Prague
  - Institut klinicke a experimentalni mediciny, Prague
  - Endohope klinika sro, Prague
  - Endokrinologie Cerny Most sro, Prague
- Denmark (6):
  - Sanos Gandrup, Gandrup
  - Gentofte Hospital, Hellerup
  - Sanos Clinic, Herlev
  - Steno Diabetes Center Copenhagen, Herlev
  - Regionshospitalet Godstrup, Herning
  - Hvidovre Hospital, Hvidovre
- Finland (3):
  - Obesity Research Unit, Helsinki
  - Health Step Finland, Kuopio
  - Oulu University Hospital, Oulu
- Germany (30):
  - Universitaetsklinikum Aachen, Aachen
  - Kardiologische Praxis Dr med Wolfgang Jungmair, Bad Homburg
  - Universitaets-Herzzentrum Freiburg - Bad Krozingen, Bad Krozingen
  - Diabetespraxis Bad Mergentheim, Bad Mergentheim
  - Universitaetsklinikum der Ruhr-Universitaet Bochum, Bad Oeynhausen
  - Charite - Universitaetsmedizin Berlin, Campus Mitte, Berlin
  - Velocity Clinical Research GmbH, Berlin
  - Diabetespraxis Dr. Hermann Braun, Berlin
  - Mvz am Bahnhof Spandau, Berlin
  - Universitaetsklinikum Dresden, Dresden
  - Zentrum fuer Klinische Studien Suedbrandenburg GmbH, Elsterwerda
  - InnoDiab Forschung, Essen
  - Praxis am Markt Dr. Bernd Becker, Essen
  - Schwerpunktpraxis fuer Diabetes, Gefaess- & Ernaehrungsmedizin, Falkensee
  - ClinPhenomics CVC GmbH, Frankfurt am Main
  - Diabeteszentrum Hamburg West, Hamburg
  - Endokrinologikum Hamburg, Hamburg
  - Diabetologische Schwerpunktpraxis Hohenmoelsen, Hohenmölsen
  - Braun Ambulantes Herzzentrum Kassel, Kassel
  - Universitaetsklinikum Leipzig, Leipzig
  - AmBeNet GmbH, Leipzig
  - Universitaetsklinikum Schleswig-Holstein - Luebeck, Lübeck
  - Marienhaus Klinikum Mainz, Mainz
  - Kardiologische Praxis Doktor Jens Taggeselle, Markkleeberg
  - Centrum für Diagnostik und Gesundheit, München
  - Zentrum fuer Diabtes und Gefaesskrankheiten im Franziskus Carré Muenster, Münster
  - Praxis Segner - Dr. Braun - Kirsch, Oberwürzbach
  - Red-Institut GmbH, Oldenburg
  - Gemeinschaftspraxis Prof Jacob/ Dr Jacob, Villingen-Schwenningen
  - Zentrum fuer klinische Forschung Allgaeu Oberschwaben, Wangen
- Italy (8):
  - IRCCS Azienda Ospedaliero Universitaria di Bologna Policlinico di Sant Orsola, Bologna
  - Universita degli Studi Gabriele D Annunzio di Chieti e Pescara, Chieti
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - IRCCS Centro Cardiologico Monzino, Milan
  - Azienda Socio Sanitaria Territoriale Fatebenefratelli Sacco, Milan
  - Ospedale Civico, Di Cristina e Benfratelli, Palermo
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Fondazione Policlinico Tor Vergata, Roma
- Japan (7):
  - Medical Corporation Hitomikai Motomachi Takatsuka Naika Clinic, Yokohama, Kanagawa
  - Doujin Memorial Foundation, Meiwa Hospital, Chiyoda-ku, Tokyo
  - Tokyo Asbo Clinic, Chuo-ku, Tokyo
  - Medical Corp Seikoukai New Medical Research System Clinic, Hachioji-shi, Tokyo
  - Medical Corporation AOT Shinagawa Strings Clinic, Minato-ku, Tokyo
  - Clinical Research Hospital Tokyo, Shinjuku-ku, Tokyo
  - Medical Corporation Hanabusakai Shinei Medical Healthcare Clinic, Suginami-ku, Tokyo
- Poland (12):
  - Gabinet Leczenia Otylosci i Chorob Dietozaleznych dr hab n med Lucyna Ostrowska, Bialystok
  - Kresmed Spolka z Ograniczona Odpowiedzialnoscia, Bialystok
  - Etg Lublin Spzoo, Dębica
  - Futuremeds Spolka z ograniczona odpowiedzialnoscia, Gdynia
  - Uniwersyteckie Centrum Kliniczne im Prof K Gibinskiego Slaskiego UM w Katowicach, Katowice
  - Salvia-Lekston i Madej Spolka Jawna, Katowice
  - Centrum Terapii Wspolczesnej J M Jasnorzewska Spolka Komandytowo Akcyjna, Lodz
  - Ekamed Spolka z Ograniczona Odpowiedzialnoscia, Lublin
  - Centrum Zdrowia Metabolicznego Pawel Bogdanski, Poznan
  - Clinical Research Center Spzoo Medic-R Spolka Komandytowa, Poznan
  - Futuremeds Spolka z ograniczona odpowiedzialnoscia, Warsaw
  - Clinical Best Solutions Sp zoo Spolka komandytowa, Warsaw
- Puerto Rico (4):
  - Ponce Medical School Foundation Inc, Ponce
  - Puerto Rico Medical Research Inc., Ponce
  - Latin Clinical Trial Center, San Juan
  - Wellness Clinical Research Vega Baja, Vega Baja
- South Korea (19):
  - Korea University Ansan Hospital, Ansan-si, Gyeonggi-do
  - Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do
  - The Catholic University of Korea Bucheon St Marys Hospital, Bucheon, Gyeonggi-do
  - Dong-A University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Yeungnam University Medical Center, Daegu
  - Daejeon Eulji Medical Center, Eulji University, Daejeon
  - Konyang University Hospital, Daejeon
  - Dongguk University Ilsan Hospital, Goyang-si, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - KyungHee University Gangdong Hospital, Seoul
  - Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul
  - The Catholic University of Korea Yeouido St Marys Hospital, Seoul
  - Ajou University Hospital, Suwon-si Gyeonggi-do
  - Pusan National University Yangsan Hospital, Yangsan-si, Gyeongsangnam-do
- Spain (11):
  - Centro Periferico de Especialidades Bola Azul, Almería, Andalusia
  - Hospital Vithas Sevilla, Castilleja de la Cuesta, Andalusia
  - Hospital Infanta Elena, Huelva, Andalusia
  - Hospital Virgen del Camino, Sanlúcar de Barrameda, Andalusia
  - Nuevas Tecnologias en Diabetes y Endocrinologia, Seville, Andalusia
  - Hospital Quironsalud Infanta Luisa, Seville, Andalusia
  - Hospital Medico Quirurgico San Rafael, A Coruña, Galicia
  - Clinica Ruber SA, Pozuelo de Alarcón, Madrid
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Clinica Juaneda, Palma
  - Hospital Universitario Doctor Peset, Valencia
- Switzerland (5):
  - Universitaetsspital Basel, Basel
  - Hopitaux Universitaires de Geneve, Geneva
  - Kantonsspital Sankt Gallen, Sankt Gallen
  - Stoffwechselzentrum Sankt Gallen, Sankt Gallen
  - Universitaetsspital Zuerich, Zurich
- United Kingdom (15):
  - Ormeau Clinical Trials Ltd, Belfast
  - FutureMeds Birmingham, Birmingham
  - Layton Medical Centre, Blackpool
  - Waterloo Medical Centre, Blackpool
  - Southmead Hospital, Bristol
  - The Rame Group Practice, Cornwall
  - Staploe Medical Centre, Ely
  - FutureMeds Glasgow, Glasgow
  - Hull Royal Infirmary, Hull
  - NIHR Leicestershire & Northamptonshire Commercial Research Delivery Centre, Leicester
  - Aintree University Hospital, Liverpool
  - FutureMeds Newcastle, Newcastle upon Tyne
  - Atlantic Medical Group, Penzance
  - Clifton Medical Centre, Rotherham
  - Ashfields Primary Care Centre, Sandbach

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com